CLINICAL TRIAL: NCT06824727
Title: Collection of Peripheral Blood From Patients With Hematologic Malignancies With Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE2424; 2R44HL145948-02 (NIH)
Record Dates: First submitted 2025-02-12; First posted 2025-02-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Thrombocytopenia
Keywords: Stem Cell Transplant
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample Collection
  Interventions: Other: Baseline cell blood counts

INTERVENTIONS:
Other: Baseline cell blood counts — Obtain one peripheral blood sample from participants who have severe thrombocytopenia defined as 30,000 platelets/mcl or less

SUMMARY:
The purpose of the research project is to collect one blood sample from participants who are affected by very low platelets as a result of their condition or their treatment.

DETAILED DESCRIPTION:
Thrombocytopenia, a condition characterized by abnormally low platelet counts, is a major complication for patients undergoing stem cell transplantation (SCT) as well as patients treated with high doses of chemotherapy for hematologic malignancies1

. Stem cell transplant is a potentially curative treatment for various blood cancers and other lifethreatening diseases. However, the conditioning regimens used before SCT, typically involving high-dose chemotherapy and/or radiation therapy, often damage the bone marrow, leading to a temporary but profound drop in platelet production. Consequences of Thrombocytopenia in SCT patients and those treated with intense chemotherapy for hematologic malignancies.

* Increased Bleeding Risk: Platelets are essential for blood clotting, and thrombocytopenia significantly increases the risk of bleeding, both minor and potentially life-threatening. This can occur anywhere in the body, including the gastrointestinal tract, lungs, and brain
* Extended Hospital Stays: Bleeding complications often require transfusions of donor platelets, which can be scarce and carry risks of transfusion reactions and infections. This can lead to prolonged hospital stays and delays in engraftment (recovery of normal blood cell production).

Current Management of Thrombocytopenia in SCT:

* Prophylactic Platelet Transfusions: To prevent bleeding, patients often receive prophylactic platelet transfusions, even if they have no symptoms. However, this approach carries risks of transfusion reactions and can strain the blood supply2
* Thrombopoietin-Stimulating Agents (TSAs): These medications stimulate the bone marrow to produce more platelets, but their effectiveness is limited and they may not be suitable for all patients3

The current protocol is aimed at testing a nanoparticle - based product that could act hemostatically as a platelet replacement. This could have several benefits.

* Addressing Platelet Shortage: The development of safe and effective off the shelf platelet replacement could address the shortage of donor platelets and reduce the reliance on donors and transfusions.
* Targeted and Controlled Platelet Function: Specific dosing studies could help understand doses of platelet replacement products for treatment of bleeding as well as the doses and concentrations required for achieve hemostasis and prevent bleeding.
* Reduced Transfusion-Related Risks: Avoiding frequent transfusions would eliminate the risk of transfusion reactions and infections, leading to improved patient safety and outcomes

This protocol is aimed at obtaining one peripheral blood sample from patients who have severe thrombocytopenia defined as 30,000 platelets/mcl or less, so that the effects of a platelet replacement product can be tested in vitro by Haima Therapeutics. This research cannot be done on samples that have been stored or frozen, as these conditions negatively impact remaining platelet function, altering the baseline of the experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older
2. Platelet counts of 30,000/mcl or less

Exclusion Criteria:

1. Chemotherapy within the last 24 hours from the planned blood sample draw for research purposes.
2. Use of anticoagulant agents in the last 48 hours.
3. Active infection (i.e. one that has received less than 48 hours of active treatment).
4. Adults 89 years or older

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be collected from participants from the bone marrow transplant inpatient service and outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Sample collection of peripheral blood from patients experiencing thrombocytopenia | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caimi, MD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided